CLINICAL TRIAL: NCT01069406
Title: The Association Between Uterine Artery Notch and First Trimester Bleeding
Status: Completed | Type: Observational
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Gali Pariente, Dr, Soroka University Medical Center
Other Study IDs: sor493710CTIL
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Uterine Artery Notch; First Trimester Bleeding
Keywords: notch; uterine; first; bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- presence of uterine artery notch: patients with uterine artery notch during the 2nd and 3rd trimester

SUMMARY:
The purpose of the present study is to evaluate the occurrence of first trimester bleeding among patients with abnormal uterine artery Doppler.

A prospective study is designed and two groups will be studied; patients with abnormal uterine artery Doppler at second trimester (study group) and patient with normal uterine artery Doppler at second trimester (control group).The patients will be asked, as part of the routine history taken before the US about having first trimester bleeding during the current pregnancy.

DETAILED DESCRIPTION:
The purpose of the present study is to evaluate the occurrence of first trimester bleeding among patients with abnormal uterine artery Doppler.

A prospective study is designed and two groups will be studied; patients with abnormal uterine artery Doppler at second trimester (study group) and patient with normal uterine artery Doppler at second trimester (control group). Both the study group and the control group represent high risk pregnant patients and the Doppler flows are done as part of the patient's predictive risk for placental associated abnormalities. The patients will be asked, as part of the routine history taken before the US about having first trimester bleeding during the current pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with abnormal uterine artery Doppler at second trimester

Exclusion Criteria:

* Multi fetal pregnancies
* Patients without known gestational age (according to last month period or first trimester ultrasound
* Pregnancies with congenital structural or chromosomal anomalies
* Lack of prenatal care

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with abnormal uterine artery Doppler at second trimester. pregnant women with eather: elevated HCG and/or aFP at triple test, patients with history of pre eclampsia, IUGR, APD, and patients with thrombophilia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Us unit, Soroka Medical Center, Beer Sheva, Israel